CLINICAL TRIAL: NCT03216057
Title: Effect of Omega-3 Fatty Acids Supplementation on Hypertriglyceridemia in Pediatric Patients With Obesity. A Randomized, Double Blind, Placebo-controlled Clinical Trial.
Brief Title: Effect of Omega-3 Fatty Acids Supplementation on Hypertriglyceridemia in Pediatric Patients With Obesity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Blanca Estela Del Rio Navarro, Principal Investigator, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIM/2008/006
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hypertriglyceridemia; Pediatric Obesity
Keywords: hypertriglyceridemia; pediatric obesity; omega 3
MeSH Terms: conditions — Hypertriglyceridemia; Pediatric Obesity | interventions — Docosahexaenoic Acids; Soybean Oil

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: The Masking intervention had made for investigation subjects and researchers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 fatty acid 3 grams per day (Experimental): Each capsule contains 400 mg of eicosapentaenoic acid and 200 mg of docosahexaenoic acid. We allocated five capsules per day, three in the morning and two at night, every 12 hours (8.00 am and 8:00 pm), therefore the subject ingest 2000 mg of eicosapentaenoic acid and 1000 mg of docosahexaenoic acid per day (3 grams of Omega 3 per day) by mouth for 12 weeks. The trademark is Omega Rx Dr.Sears Zone labs Inc.
  Interventions: Dietary Supplement: Omega-3 fatty acid 3 grams per day
- Placebo (Placebo Comparator): Each capsule contains 600 mg of soybean oil. We allocated five capsules per day, three in the morning and two at night, every 12 hours (8.00 am and 8:00 pm), therefore the subject ingest 3000 mg of soybean oil per day (3 gr soya oil per day) by mouth for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid 3 grams per day — Each capsule contains 400 mg of eicosapentaenoic acid and 200 mg of docosahexaenoic acid. We allocated five capsules per day, three in the morning and two at night, every 12 hours (8.00 am and 8:00 pm), therefore the subject ingest 2000 mg of eicosapentaenoic acid and 1000 mg of docosahexaenoic acid per day (3 gr of Omega 3 per day) by mouth for 12 weeks. The trademark is Omega RX Dr.Sears Zone labs Inc.
  Other Names: Omega-3
  Arms: Omega-3 fatty acid 3 grams per day
Dietary Supplement: Placebo — Placebo Comparator: Placebo Each capsule contains 600 mg of soybean oil. We allocated five capsules per day, three in the morning and two at night, every 12 hours (8.00 am and 8:00 pm), therefore the subject ingest 3000 mg of soybean oil per day (3 gr soya oil per day) by mouth for 12 weeks.
  Other Names: Soybean oil
  Arms: Placebo

SUMMARY:
The primary objective was to evaluate the safety and efficacy the 3 grams per day of omega-3 in adolescents with obesity and hypertriglyceridemia ( ≥ 150 mg/dl and ≤ 1000 mg/dl) for 12 weeks, compared with placebo. Half of subjects received 3 grams of omega 3, while the other half received placebo.

DETAILED DESCRIPTION:
First of all, the omega-3 free fatty acids have an important effect for lowering triglycerides through three potential mechanisms such as:

Inhibition of triacylglycerol synthesis as direct inhibition of diacyl glycerol acetyl transferase and phosphatidic acid phosphohydrolase results in lowering triacylglycerol production.

Simulation of fatty acid oxidation through activation of peroxisome proliferation activated receptor stimulates hepatic mitochondrial and peroxisomal beta oxidation of fatty acids. Decreased availability of fatty acids for triacylglycerol synthesis results in lowering plasma triacylglycerol levels Lipoprotein Lipase mediated clearance. One of the first randomized double blind placebo controlled clinical trials was managed by Harris in 1997 in adult subjects with an average age of 46 ± 11 years and severe hypertriglyceridemia (500-2000 mg / dl) 20 subjects received placebo and 22 subjects 4 grams of omega-3. The mean percent change from baseline in the omega-3 group was -45 ± 23% and in the placebo group was -16 ± 35% (p <0.0001).

Also, more clinical trials have recently been conducted with similar results such as the most recent randomized, double-blind, placebo-controlled clinical trial that was conducted by Ta-Chen Su in Taiwan in adults with hypertriglyceridemia (200-1000 mg / dl). The first group received 4 grams of omega-3 (n = 84), the second group received 2 grams of omega-3 (n = 82) and the third group received placebo (n = 87). The mean percent change from baseline in the 4 grams of omega-3 group was -32.1%, in the 2 grams group of omega-3 was -29.7% and in the placebo group was -5.4% (p <0.0001) What is more, the strongest scientific evidence in favor of supplementation of omega-3 acids fatty was determined by two meta-analysis, the first study was published by Harris in 1997 that included 72 placebo-controlled clinical trials, the study showed a reduction of 25-30% triglycerides levels with doses of 3-4 g omega-3 compared with placebo in subjects with triglycerides levels ≥500mg / dl. The second meta-analysis by Balk that included 17 clinical trials (7,803 patients) with different doses of omega-3 (0.8-5.4 g). The net reduction in triglycerides levels was -27 mg / dl (IC95% 22-30), p <0.0001 In addition, the American Heart Association based on the meta-analysis by Harris currently recommends the administration of 2 to 4 grams of omega-3 per day for the treatment of severe hypertriglyceridemia (≥500mg / dl) in adult patients.

Secondly, the Task Force for the Management of Dyslipidaemias of the European Society of Cardiology (ESC) and European Atherosclerosis Society (EAS) currently recommends that if hypertriglyceridemia is not able to reduce with statins or fibrates the physician will prescribe 2-4 grams of omega-3 fatty acids to reduce triglyceride levels in adult patients.

Finally, the Food Drug Administration (FDA) in 2004 authorized the administration of 2 to 4 grams of omega-3 per day for the treatment of severe hypertriglyceridemia (≥500mg / dl) in adult patients.

There is enough evidence that medical literature supports the use of omega-3 in adult patients for treatment of hypertriglyceridemia even the American Heart Association has made the recommendation in its Scientific Statement but unfortunately in children the information about the use of omega-3 for hypertriglyceridemia is insufficient to make clinical decisions.

There are no specific recommendations and dosages of omega-3 in children and adolescents for the treatment of hypertriglyceridemia.

A randomized, double-blind placebo controlled clinical trials are necessary to assess the efficacy and safety of omega-3 fatty acids for the treatment of hypertriglyceridemia in children and adolescents.

Main objective:

Assessing the efficacy and safety of supplementation of 3 grams of omega-3 fatty acids for 12 weeks on serum triglycerides in adolescents with obesity and hypertriglyceridemia compared to a control group that received placebo.

Secondary objective:

Assessing the efficacy and safety of supplementation of 3 grams of omega-3 fatty acids for 12 weeks on serum cholesterol, HDL-C, glucose and uric acid in adolescents with obesity and hypertriglyceridemia compared to a control group that received placebo.

Study plan detailing the procedures.

Visit 1 Enrollment:

The subject was picked up by the Allergy Department and Obesity Clinic. Informed consent and informed assent. Demography (date of birth, gender) and evaluation of Inclusion/Exclusion criteria Medical. Surgical history physical examination and anthropometry (weight, height, body mass index, abdominal perimeter, waist and hip). Pulse and blood pressure. Pregnancy test. Fasting venous blood samples of 12 hours for the measurement of triglycerides and metabolic profile. Food recommendation was indicated by the Pediatric Clinical Nutrition Service. Physical activity was indicated with a 30-minute walk per day for seven days per week by the Pediatric Clinical Nutrition service.

Visit 2 Randomization:

Triglyceride levels were reviewed, in case of report ≥150 mg / dl and ≤ 1000 mg/dl the subjects were randomized.

The type of randomization used was blocked randomisation, number of subjects per block were 10 and number of blocks were 13. (130 subjects were randomized).

Allocation of omega-3 or placebo capsules for all randomized subjects and beginning of the week 0 of treatment.

Visit 3 Treatment week 4 Allocation of omega-3 or placebo capsules. Checking of adverse effects. Accounting of capsules. Supervision of compliance diary of omega-3 or placebo capsules. Supervision of compliance diary food recommendation. Supervision of compliance physical activity

Visit 4 Treatment week 8 Allocation of omega-3 or placebo capsules. Checking of adverse effects. Accounting of capsules. Supervision of compliance diary of omega-3 or placebo capsules. Supervision of compliance diary food recommendation. Supervision of compliance physical activity.

Visit 5 Treatment week 12 Checking of adverse effects. Accounting of capsules. Supervision of compliance diary of omega-3 or placebo capsules. Supervision of compliance diary food recommendation. Supervision of compliance physical activity.

Follow-up telephone call week 16. A follow-up telephone was performed 4 weeks after the visit 5. At the follow-up telephone call, the investigator checked adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10-16 years old
* Informed consent from a parent or legal guardian of minors or adult subject
* Written assent from the adolescent to participate in the study
* Obese patients (Body Mass Index ≥95th percentile according to the National Center for Health Statistics, Center for Disease Control and Prevention [CDC].
* Fasting Serum triglycerides ≥150 mg/dL and ≤1000 mg/dL.
* Cooperation to ingest capsules (omega-3 or placebo) and taking laboratories

Exclusion Criteria:

* The subjects must not had received pharmacology treatment for hypertriglyceridemia six months before and at the time of enrollment.
* Treatment with medications that affect triglyceride levels, including oral hypoglycemic agents or insulin.
* Pregnancy or positive urine pregnancy test for those females who have begun menstruating.
* Known Bleeding Disorder or Coagulopathy or treatment with anticoagulant medications or low platelet counts, abnormal PT, or PTT.
* Subjects with mental delayed.
* Neurological disorder.
* Subjects with Cardiopathy
* Subjects with gastroesophageal reflux
* Endocrinopathies such as thyroid disorder, Hypothalamic disorder and Type 1 or 2 diabetes or fasting glucose that is >=126 mg/dl.
* Subjects with liver disease
* Familial hypertriglyceridemia.
* Familial hypercholesterolemia
* Polycystic ovary syndrome
* Use of contraceptives by any way of administration 6 months before and at the time of enrollment.
* Use of vitamins 6 months before and at the time of enrollment.
* Allergy to fish oil.
* Allergy to soybean oil.

Elimination criteria:

* Subject or parents´ subject either decision to discontinue of the study at any time without prejudice to further treatment.
* Serious adverse event.
* Safety reason as judged by the investigator.
* Pregnancy.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2008-05-20 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harris WS, Ginsberg HN, Arunakul N, Shachter NS, Windsor SL, Adams M, Berglund L, Osmundsen K. Safety and efficacy of Omacor in severe hypertriglyceridemia. J Cardiovasc Risk. 1997 Oct-Dec;4(5-6):385-91. PMID 9865671
- [Result] Harris WS. n-3 fatty acids and serum lipoproteins: human studies. Am J Clin Nutr. 1997 May;65(5 Suppl):1645S-1654S. doi: 10.1093/ajcn/65.5.1645S. PMID 9129504
- [Result] Jacobson TA. Role of n-3 fatty acids in the treatment of hypertriglyceridemia and cardiovascular disease. Am J Clin Nutr. 2008 Jun;87(6):1981S-90S. doi: 10.1093/ajcn/87.6.1981S. PMID 18541599
- [Result] Miller M, Stone NJ, Ballantyne C, Bittner V, Criqui MH, Ginsberg HN, Goldberg AC, Howard WJ, Jacobson MS, Kris-Etherton PM, Lennie TA, Levi M, Mazzone T, Pennathur S; American Heart Association Clinical Lipidology, Thrombosis, and Prevention Committee of the Council on Nutrition, Physical Activity, and Metabolism; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease. Triglycerides and cardiovascular disease: a scientific statement from the American Heart Association. Circulation. 2011 May 24;123(20):2292-333. doi: 10.1161/CIR.0b013e3182160726. Epub 2011 Apr 18. No abstract available. PMID 21502576
- [Result] Su TC, Hwang JJ, Huang KC, Chiang FT, Chien KL, Wang KY, Charng MJ, Tsai WC, Lin LY, Vige R, Olivar JE, Tseng CD. A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Assess the Efficacy and Safety of Ethyl-Ester Omega-3 Fatty Acid in Taiwanese Hypertriglyceridemic Patients. J Atheroscler Thromb. 2017 Mar 1;24(3):275-289. doi: 10.5551/jat.34231. Epub 2016 Sep 6. PMID 27600795
- [Result] Kastelein JJ, Maki KC, Susekov A, Ezhov M, Nordestgaard BG, Machielse BN, Kling D, Davidson MH. Omega-3 free fatty acids for the treatment of severe hypertriglyceridemia: the EpanoVa fOr Lowering Very high triglyceridEs (EVOLVE) trial. J Clin Lipidol. 2014 Jan-Feb;8(1):94-106. doi: 10.1016/j.jacl.2013.10.003. Epub 2013 Oct 14. PMID 24528690
- [Result] Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Z, Riccardi G, Taskinen MR, Tokgozoglu L, Verschuren WM, Vlachopoulos C, Wood DA, Zamorano JL. [2016 ESC/EAS Guidelines for the Management of Dyslipidaemias]. Kardiol Pol. 2016;74(11):1234-1318. doi: 10.5603/KP.2016.0157. No abstract available. Polish. PMID 27910077
- [Result] Balk EM, Lichtenstein AH, Chung M, Kupelnick B, Chew P, Lau J. Effects of omega-3 fatty acids on serum markers of cardiovascular disease risk: a systematic review. Atherosclerosis. 2006 Nov;189(1):19-30. doi: 10.1016/j.atherosclerosis.2006.02.012. Epub 2006 Mar 10. PMID 16530201
- [Result] Bays HE, Tighe AP, Sadovsky R, Davidson MH. Prescription omega-3 fatty acids and their lipid effects: physiologic mechanisms of action and clinical implications. Expert Rev Cardiovasc Ther. 2008 Mar;6(3):391-409. doi: 10.1586/14779072.6.3.391. PMID 18327998
- [Result] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2889-934. doi: 10.1016/j.jacc.2013.11.002. Epub 2013 Nov 12. No abstract available. PMID 24239923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were enrolled from Obesity Clinic and Department of Pediatric Allergy and Clinical Immunology of the Children's Hospital of Mexico.
Pre-assignment Details: First of all, the researcher has enrolled 168 subjects, who were assessed for eligibility, but 38 subjects have done screen failure because they have not met all the inclusion criteria, therefore only 130 subjects, who have started the study, were randomized.
Groups:
- Omega-3: Each capsule contains 400 mg of eicosapentaenoic acid and 200 mg of docosahexaenoic acid. We allocated five capsules per day, three in the morning and two at night, every 12 hours (8.00 am and 8:00 pm), therefore the subject ingest 2000 mg of eicosapentaenoic acid and 1000 mg of docosahexaenoic acid per day (3 grams of Omega 3 per day) by mouth for 12 weeks. The trademark is Omega Rx Dr.Sears Zone labs Inc.
  Omega-3 fatty acid 3 grams per day: Each capsule contains 400 mg of eicosapentaenoic acid and 200 mg of docosahexaenoic acid. We allocated five capsules per day, three in the morning and two at night, every 12 hours (8.00 am and 8:00 pm), therefore the subject ingest 2000 mg of eicosapentaenoic acid and 1000 mg of docosahexaenoic acid per day (3 gr of Omega 3 per day) by mouth for 12 weeks. The trademark is Omega RX Dr.Sears Zone labs Inc.
Period: Overall Study
Arm/Group | Omega-3 | Placebo
Started | 65 | 65
Completed | 63 | 63
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 | Placebo | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (1.6) | 12.5 (1.5) | 12.3 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 42 | 80
  Male | 27 | 23 | 50
Weight [Mean (Standard Deviation); unit: Kilograms] | 70.4 (16.2) | 68.4 (14.2) | 69.4 (15.2)
Height [Mean (Standard Deviation); unit: centimeters] | 155.0 (10.7) | 154.5 (10.7) | 154.8 (10.7)
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 28.9 (3.8) | 28.2 (3.0) | 28.6 (3.4)
Abdominal circumference [Mean (Standard Deviation); unit: centimeters] | 95.5 (10.6) | 93.5 (8.4) | 94.5 (9.6)
Hip circumference [Mean (Standard Deviation); unit: centimeters] | 91.6 (10.0) | 90.1 (7.5) | 90.8 (8.8)
Waist circumference [Mean (Standard Deviation); unit: centimeters] | 99.8 (11.05) | 98.9 (8.6) | 99.4 (9.8)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 222.1 (62.3) | 222.6 (75.9) | 222.4 (69.2)
Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 165.0 (30.2) | 157.9 (38.3) | 161.4 (34.5)
Glucose [Mean (Standard Deviation); unit: mg/dl] | 86.9 (8.7) | 85.3 (13.1) | 86.1 (11.1)
HDL-C [Mean (Standard Deviation); unit: mg/dl] | 34.6 (9.8) | 32.6 (6.7) | 33.6 (8.4)
Uric acid [Mean (Standard Deviation); unit: mg/dl] | 6.0 (1.3) | 5.8 (1.0) | 5.9 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Serum Triglyceride Levels From Baseline to Week 12 of Study Treatment
Description: Percentage change in serum triglyceride levels from baseline to week 12 of study treatment
Time Frame: 12 weeks
Population: Intention to treat population (All subjects who received at least one dose of intervention were assessed in statistical analysis)
Measure: Mean (Standard Deviation); unit: Percent change (%)
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 65 | 65
Percent change (%) | -39.1 (24.7) | -14.6 (21.8)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Test type: Superiority — The sample size was calculated that 130 subjects randomized in a 1:1 fashion between the 2 arms have 85% power to detect a difference of at least 20% in triglyceride percentage changes compared with placebo at week 12, assuming a common standard deviation in percentage change of 35%, a 2-sided α = 0.05, and we add 20% for lost follow-up, finally the number of subjects for each arm was 65; p < 0.01, t-test, 2 sided; Mean Difference (Net) = -24.5, 95% CI 2-sided [-32.7 to -16.2]

2. Primary Outcome: Milligram Change in Serum Triglyceride Levels From Baseline to Week 12 of Study Treatment
Description: Milligram Change in Serum Triglyceride Levels From Baseline to Week 12 of Study Treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 65 | 65
mg/dl | 127.7 (45.5) | 187.6 (80.4)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Test type: Superiority; p < 0.01, t-test, 2 sided; Mean Difference (Net) = -59.9, 95% CI 2-sided [-83.0 to -36.8]

3. Secondary Outcome: Percentage Change in Serum Cholesterol Levels From Baseline to Week 12 of Study Treatment
Description: Percentage Change in Serum Cholesterol Levels From Baseline to Week 12 of Study Treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percent change (%)
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 65 | 65
Percent change (%) | -2.9 (19.5) | 6.1 (20.6)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = -9.0, 95% CI 2-sided [-16.1 to -1.9]

4. Secondary Outcome: Milligram Change in Serum Cholesterol Levels From Baseline to Week 12 of Study Treatment
Description: Milligram Change in Serum Cholesterol Levels From Baseline to Week 12 of Study Treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 65 | 65
mg/dl | 157.4 (31.4) | 162.4 (30.7)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Test type: Superiority; p = 0.3, t-test, 2 sided; Mean Difference (Net) = -4.9, 95% CI 2-sided [-15.8 to 6.05]

5. Secondary Outcome: Percentage Change in Serum HDL-C Levels From Baseline to Week 12 of Study Treatment
Description: Percentage Change in Serum HDL-C Levels From Baseline to Week 12 of Study Treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percent change (%)
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 65 | 65
Percent change (%) | 3.8 (22.3) | 16.2 (27.5)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Test type: Superiority; p < 0.01, t-test, 2 sided; Mean Difference (Net) = -12.4, 95% CI 2-sided [-21.2 to -3.5]

6. Secondary Outcome: Milligram Change in Serum HDL-C Levels From Baseline to Week 12 of Study Treatment
Description: Milligram Change in Serum HDL-C Levels From Baseline to Week 12 of Study Treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 65 | 65
mg/dl | 34.4 (5.2) | 36.7 (5.8)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Net) = -2.2, 95% CI 2-sided [-4.1 to -0.3]

7. Secondary Outcome: Percentage Change in Serum Glucose Levels From Baseline to Week 12 of Study Treatment
Description: Percentage Change in Serum Glucose Levels From Baseline to Week 12 of Study Treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percent change (%)
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 65 | 65
Percent change (%) | -0.4 (10.1) | 0.7 (17.7)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Test type: Superiority; p = 0.6, t-test, 2 sided; Mean Difference (Net) = -1.2, 95% CI 2-sided [-6.3 to 3.8]

8. Secondary Outcome: Milligram Change in Glucose Levels From Baseline to Week 12 of Study Treatment
Description: Milligram Change in Glucose Levels From Baseline to Week 12 of Study Treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 65 | 65
mg/dl | 86.1 (8.6) | 84.1 (7.9)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Test type: Superiority; p = 0.1, t-test, 2 sided; Mean Difference (Net) = 1.9, 95% CI 2-sided [-0.9 to 4.9]

9. Secondary Outcome: Percentage Change in Serum Uric Acid Levels From Baseline to Week 12 of Study Treatment
Description: Percentage Change in Serum Uric Acid Levels From Baseline to Week 12 of Study Treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percent change (%)
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 65 | 65
Percent change (%) | -1.9 (26.0) | -15.3 (16.0)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Test type: Superiority; p < 0.01, t-test, 2 sided; Mean Difference (Net) = 13.4, 95% CI 2-sided [5.8 to 21]

10. Secondary Outcome: Milligram Change in Serum Uric Acid Levels From Baseline to Week 12 of Study Treatment
Description: Milligram Change in Serum Uric Acid Levels From Baseline to Week 12 of Study Treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 65 | 65
mg/dl | 5.7 (1.4) | 4.8 (0.8)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Test type: Superiority; p < 0.01, t-test, 2 sided; Mean Difference (Net) = 0.8, 95% CI 2-sided [0.4 to 1.2]

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Placebo: Each capsule contains 600 mg of soybean oil. We allocated five capsules per day, three in the morning and two at night, every 12 hours (8.00 am and 8:00 pm), therefore the subject ingest 3000 mg of soybean oil per day (3 gr soya oil per day) by mouth for 12 weeks.
  Placebo: Placebo Comparator: Placebo. Each capsule contains 600 mg of soybean oil. We allocated five capsules per day, three in the morning and two at night, every 12 hours (8.00 am and 8:00 pm), therefore the subject ingest 3000 mg of soybean oil per day (3 gr soya oil per day) by mouth for 12 weeks.
Arm/Group | Omega-3 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 27/65 | 4/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omega-3 (N=65) | Placebo (N=65)
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Fish taste belch (Gastrointestinal disorders) | 18 | 0
Nausea (Gastrointestinal disorders) | 5 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes